CLINICAL TRIAL: NCT04590326
Title: A Phase 1/2 Study of REGN5668 (MUC16xCD28, a Costimulatory Bispecific Antibody) Administered in Combination With Other Agents in MUC16 + Malignancies
Brief Title: A Study to Find Out How Safe REGN5668 is and How Well it Works In Adult Women When Given With Either Cemiplimab, or Cemiplimab + Fianlimab, or Ubamatamab
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5668-ONC-1938; 2022-501904-83-00 (EU CTIS Number)
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Endometrial Cancer
Keywords: Progressive; Recurrent; Refractory; Serum CA-125 levels >= 2x ULN
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Recurrence | interventions — cemiplimab; sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1 (Experimental): REGN5668 in combination with cemiplimab, or cemiplimab + fianlimab
  Interventions: Drug: REGN5668; Drug: Cemiplimab; Drug: Cemiplimab + Fianlimab [Fixed Dose Combination (FDC)]
- Module 2 (Experimental): REGN5668 and ubamatamab
  Interventions: Drug: REGN5668; Drug: Ubamatamab; Drug: Sarilumab

INTERVENTIONS:
Drug: REGN5668 — Administer per the protocol
Drug: Cemiplimab — Administer per the protocol
  Other Names: REGN2810; Libtayo®
  Arms: Module 1
Drug: Ubamatamab — Administer per the protocol
  Other Names: REGN4018
  Arms: Module 2
Drug: Sarilumab — Administer per the protocol
  Other Names: Kevzara®
  Arms: Module 2
Drug: Cemiplimab + Fianlimab [Fixed Dose Combination (FDC)] — Administer per the protocol
  Arms: Module 1

SUMMARY:
This study is researching an investigational drug called REGN5668 :

* alone or,
* combined with cemiplimab (also known as REGN2810) or,
* combined with both cemiplimab and fianlimab (also known as REGN3767), or
* combined with ubamatamab (also known as REGN4018), with or without sarilumab.

The main purposes of this study are to:

* Learn about the safety and profile of any side effects from the study drugs and to determine the highest, safe dose that can be given to participants with ovarian cancer or cancer of the uterus
* Look for signs that the study drugs can treat ovarian cancer or cancer of the uterus

This study has 2 parts. The purpose of Part 1 (Escalation) is to find the highest, safe dose of the study drug(s). The purpose of Part 2 (Expansion) is to use the doses chosen in Part 1. Participants with cancer of the uterus will only participate in Part 2.

The study is looking at several other research questions, including:

* Side effects that may be experienced by participants taking REGN5668 alone and/or in combination with cemiplimab, cemiplimab and fianlimab, or ubamatamab
* How REGN5668 works in the body either alone and/or in combination with cemiplimab, cemiplimab and fianlimab, or ubamatamab
* How much of the study drugs (REGN5668, cemiplimab, fianlimab, ubamatamab) are in the blood
* To see if REGN5668 in combination with cemiplimab, cemiplimab and fianlimab, or ubamatamab works to treat cancer

ELIGIBILITY:
Key Inclusion Criteria:

1. Ovarian Cancer Cohorts Only: Has histologically or cytologically confirmed diagnosis of advanced epithelial ovarian cancer (except carcinosarcoma), primary peritoneal, or fallopian tube cancer that has received at least 1 line of platinum-based systemic therapy as defined in the protocol
2. Expansion cohorts only: Has at least 1 lesion that is measurable by RECIST 1.1 as described in the protocol.
3. Has a serum CA-125 level ≥2x ULN (in screening, not applicable to endometrial cohorts)
4. Has adequate organ and bone marrow function as defined in the protocol
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Has a life expectancy of at least 3 months
7. Endometrial Cancer Cohorts Only: histologically confirmed endometrial cancer that has progressed or recurrent after prior anti-PD-1 therapy and platinum-based chemotherapy as described in the protocol

Key Exclusion Criteria:

1. Current or recent (as defined in the protocol) treatment with an investigational agent, systemic biologic therapy, or anti-cancer immunotherapy
2. Has had another malignancy within the last 5 years that is progressing, requires active treatment, or has a high likelihood of recurrence as defined in the protocol
3. Prior treatment with a Mucin 16 (MUC16)-targeted therapy
4. Ovarian Expansion cohorts only: More than 5 prior lines of systemic therapy
5. Has any condition that requires ongoing/continuous corticosteroid therapy as defined in the protocol within 1 week prior to the first dose of study drug
6. Has ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments as defined in the protocol
7. Has untreated or active primary brain tumor, CNS metastases, leptomeningeal disease, or spinal cord compression as defined in the protocol
8. Has history of clinically significant cardiovascular disease as defined in the protocol
9. Has known allergy or hypersensitivity to cemiplimab and/or components of study drug(s).

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | 42 days
  Dose escalation phase, Module 1
Incidence of DLTs | 21 days post combination administration
  Dose escalation phase, Module 2
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Through study completion, up to 5 years
  Primary: Dose escalation phase Secondary: Dose expansion phase
Incidence of Serious Adverse Events (SAEs) | Through study completion, up to 5 years
  Primary: Dose escalation phase Secondary: Dose expansion phase
Incidence of deaths | Through study completion, up to 5 years
  Primary: Dose escalation phase Secondary: Dose expansion phase
Incidence of laboratory abnormalities (Grade 3 or higher per National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0 [v5.0]) | Through study completion, up to 5 years
  Primary: Dose escalation phase Secondary: Dose expansion phase
Concentrations of REGN5668 in serum when dosed alone and in combination with cemiplimab or ubamatamab | Through study completion, up to 5 years
  Primary: Dose escalation phase
Objective Response Rate (ORR) defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Eisenhauer, 2009) of REGN5668 in combination with cemiplimab, cemiplimab + fianlimab, or ubamatamab (separately by cohort and combination) | Through study completion, up to 5 years
  Primary: Dose expansion phase

SECONDARY OUTCOMES:
ORR based on RECIST 1.1 | Through study completion, up to 5 years
  Dose escalation phase
Best Overall Response (BOR) based on RECIST 1.1 | Through study completion, up to 5 years
  Dose escalation and expansion phases
Duration Of Response (DOR) based on RECIST 1.1 | Through study completion, up to 5 years
  Dose escalation and expansion phases
Disease Control Rate (DCR) based on RECIST 1.1 | Through study completion, up to 5 years
  Dose escalation and expansion phases
Progression-Free Survival (PFS) based on RECIST 1.1 | Through study completion, up to 5 years
  Dose escalation and expansion phases
Cancer Antigen 125 (CA-125) change from baseline after treatment with REGN5668 in combinations with cemiplimab, cemiplimab + fianlimab, or ubamatamab (separately by cohort and combination) | Through study completion, up to 5 years
  Dose escalation and expansion phases
Concentration of REGN5668 in serum over time when dosed alone and in combination with cemiplimab, cemiplimab + fianlimab, or ubamatamab | Through study completion, up to 5 years
  Dose escalation and expansion phases
Presence or absence of anti-drug antibodies against REGN5668 | Through study completion, up to 5 years
  Dose escalation and expansion phases
Presence or absence of anti-drug antibodies against ubamatamab | Through study completion, up to 5 years
  Dose escalation and expansion phases
Presence or absence of anti-drug antibodies against cemiplimab | Through study completion, up to 5 years
  Dose escalation and expansion phases
Presence or absence of anti-drug antibodies against fianlimab | Through study completion, up to 5 years
  Dose escalation and expansion phases

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (24):
- United States (13):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - The City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute Brookline Avenue, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Perelman School of Medicine at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Seattle Cancer Care Alliance at South Lake Union - G3630, Seattle, Washington
- Universitair Ziekenhuis Leuven, Leuven, Vlaams-Brabant, Belgium
- France (5):
  - Hopital Lyon Sud, Pierre-Bénite, Auvergne-Rhône
  - Centre Georges Francois Leclerc, Dijon, Bourgogne-Franche-Comté
  - Centre Francois Baclesse (CFB), Caen, Normandy
  - Institut Bergonie, Bordeaux, Nouvelle-Aquitaine
  - Institut Gustave Roussy, Villejuif
- Spain (5):
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, A Coruna
  - Institut Catala dOncologia Girona, Girona
  - Ciudad Universitaria, Madrid
  - Hospital Universitario Fundacion Jimenez, Madrid
  - Hospital Universitario 12 de Octubre Universidad Complutense de Madrid UCM, Madrid

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/